CLINICAL TRIAL: NCT06439394
Title: Patient Experience Study Evaluating Effect of OM3 on Dry Eye Symptoms and Quality of Life in Patients With Mild to Moderate Dry Eye Disease
Brief Title: An Observational Study to Assess Optive MEGA-3 (OM3) on Dry Eye Symptoms and Quality of Life of Adult Participants With Mild to Moderate Dry Eye Disease (DED)
Status: Completed | Type: Observational
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Other Study IDs: P25-006
Record Dates: First submitted 2024-05-28; First posted 2024-06-03 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Dry Eye
Keywords: Dry Eye; OM3; Optive MEGA-3; AGN-OMEGA3
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- OM3: Participants will receive 1 drop of OM3 on Day 1. After Day 1, participants will administer 1-2 eye drops in each eye at least twice a day but as much as needed through Day 15.
  Interventions: Drug: Optive MEGA-3 (OM3)

INTERVENTIONS:
Drug: Optive MEGA-3 (OM3) — Eye Drops
  Other Names: Refresh MEGA-3

SUMMARY:
Dry Eye Disease (DED) is a condition where the tear film of the eye becomes unstable and along with ocular surface inflammation and damage leads to inadequate tear production and eye lubrication. This study will evaluate real-world experiences with Optive MEGA-3 (OM3) on relieving dry eye symptoms in adult participants with DED.

OM3 is an over the counter (OTC) monograph drug indicated for the temporary relief of symptoms of eye dryness. Participants will administer 1 drop of OM3 on Day 1 for the acute phase of the study, then participants will administer 1-2 eye drops in each eye at least twice a day but as much as needed through Day 15. Around 50 adult participants will be enrolled at one site in the United States.

There is expected to be no additional burden for participants in this trial. Study visits may be conducted on-site as per standard of care.

ELIGIBILITY:
Inclusion Criteria:

* During a routine visit, investigator will decide whether artificial tears are the appropriate treatment for potential participants with dry eyes and will then consider enrollment into this study.
* Participant has at least one of the following signs of dry eye:

  * Three consecutive tear break-up time (TBUT) tests <= 10 seconds in at least one eye at Screening Visit OR;
  * Grade 1 to 4 (modified National Eye Institute [NEI] Grid, score range = 0 to 5) staining in at least 1 area of the cornea (5 areas examined) or conjunctiva (6 areas examined) that is related to dry eye in at least 1 eye at Screening Visit.

Exclusion Criteria:

* Use of artificial tears in the last 24 hours.
* Use of more than 4 drops of artificial tears per day in each eye.
* Use of dry eye treatment other than artificial tears.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult participants with dry eye disease who are eligible based on the inclusion and exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2024-06-17 (Actual); Primary Completion 2024-07-18 (Actual); Study Completion 2024-07-18 (Actual)

PRIMARY OUTCOMES:
Acute Phase: Change from Baseline in Current Symptom Scores | Day 1; Hour 8
  The Current Symptom Survey is a 5-item questionnaire where the participants rate their ocular symptoms at the current moment using a scale ranging from '0 = strongly disagree' to '100 = strongly agree.'
Chronic Phase: Change from Baseline in Ocular Surface Disease Index (OSDI) Score | Day 15
  The OSDI is a 12-question survey for patients to document their dry eye disease symptoms. The OSDI consists of a 5-point scale (0=none of the time to 4=all of the time), with higher scores representing greater disability. The scores are totaled over the 12 questions and converted to a score of 0-100 (0=no disability to 100=complete disability). A negative number change from baseline represents an improvement.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (1):
- Southern College of Optometry /ID# 262668, Memphis, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Clinical Study Report Synopsis — https://www.abbvieclinicaltrials.com/study/?id=P25-006#additional-resources-section